CLINICAL TRIAL: NCT02145039
Title: Reduced Intensity Conditioning (RIC) and Transplantation of HLA(Human Leukocyte Antigen)-Haploidentical Related Bone Marrow (Haplo-BM) For Patients With Hematologic Diseases
Brief Title: Reduced Intensity Conditioning and Haploidentical Related Bone Marrow for Patients With Hematologic Diseases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Replaced by another study.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013OC116; MT2013-33C (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Acute Leukemias; Burkitt's Lymphoma; Chronic Myelogenous Leukemia
Keywords: Acute Lymphoblastic Leukemia (ALL); Acute Myelogenous Leukemia (AML); Burkitt's lymphoma; Natural killer cell malignancies; Chronic myelogenous leukemia; Myelodysplastic syndrome; Large-cell lymphoma; Hodgkin lymphoma; Multiple myeloma; Chronic lymphocytic leukemia (CLL); Small lymphocytic lymphoma (SLL); Marginal zone B-cell lymphoma; Follicular lymphoma; Lymphoplasmacytic lymphoma; Mantle-cell lymphoma; Prolymphocytic leukemia; Refractory leukemia; Myelodysplastic syndrome (MDS); Bone marrow failure syndromes; Myeloproliferative syndromes
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Dendritic Cell Sarcoma, Interdigitating; Hodgkin Disease; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Prolymphocytic; Leukemia; Bone Marrow Failure Disorders | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haploidentical stem cell transplant (Experimental): This is a treatment guideline for HLA-Haploidentical hematopoietic stem cell transplant (HSCT) using a reduced intensity conditioning (RIC) regimen. This regimen consists of fludarabine, cyclophosphamide and low dose total body irradiation (TBI).
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Biological: Haploidentical stem cell transplant

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2 IV over 30-60 minutes on days -6 through -2 before transplant.
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide 14.5 mg/kg IV over 1-2 hours on days -6 and -5 before transplant and Cyclophosphamide 50 mg/kg IV on days 3 and 4 post-transplant.
Radiation: Total Body Irradiation — TBI 200cGy on day -1 before transplant.
  Other Names: TBI
Biological: Haploidentical stem cell transplant — Non-T-cell depleted bone marrow infusion
  Other Names: HSCT

SUMMARY:
This is a treatment guideline for HLA-Haploidentical hematopoietic stem cell transplant (HSCT) using a reduced intensity conditioning (RIC) regimen. This regimen, consisting of fludarabine, cyclophosphamide and low dose total body irradiation (TBI), is designed for the treatment of patients with advanced and/or high risk diseases.

ELIGIBILITY:
Inclusion Criteria:

* Must be <75 years old with no 7/8 or 8/8 HLA-matched sibling donor
* One or more potential related mismatched donors (e.g. biologic parent (s) or siblings (full or half) or children). Low resolution using DNA based typing at HLA-A, -B and -DRB1 for potential haploidentical donors is required.
* All diseases listed below are advanced hematologic malignancies not curable by conventional chemotherapy. Responses to conventional treatment range from zero to 30% but are typically short lived.

  * Acute Lymphoblastic Leukemia (ALL) in first complete remission (CR1) that is NOT considered favorable-risk.
  * Acute Myelogenous Leukemia (AML) in first complete remission (CR1) that is NOT considered as favorable-risk.
  * Acute Leukemias in 2nd or subsequent CR
  * Biphenotypic/Undifferentiated/Prolymphocytic Leukemias in first or subsequent CR, adult T-cell leukemia/lymphoma in first or subsequent CR
  * Burkitt's lymphoma in CR2 or subsequent CR
  * Natural killer cell malignancies after response to initial therapy
  * Chronic myelogenous leukemia: all types except refractory blast crisis.
  * Large-cell lymphoma, Hodgkin lymphoma and multiple myeloma with chemotherapy sensitive disease that has failed or patients who are ineligible for an autologous transplant.
  * Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma, follicular lymphoma, which have progressed within 12 months of achieving a partial or complete remission.
  * Lymphoplasmacytic lymphoma, mantle-cell lymphoma, prolymphocytic leukemia are eligible after initial therapy if chemotherapy sensitive.
  * Refractory leukemia or MDS These patients may be taken to transplant in aplasia after induction or re-induction chemotherapy or radiolabeled antibody.
  * Bone marrow failure syndromes, except for Fanconi Anemia
  * Myeloproliferative syndromes
* Adequate organ function is defined as:

  * Cardiac: Absence of decompensated congestive heart failure, or uncontrolled arrhythmia and left ventricular ejection fraction > 35%. For children that are not able to cooperate with multigated acquisition scan (MUGA) and echocardiography, such should be clearly stated in the physician's note
  * Pulmonary: Diffusing capacity of lung for carbon monoxide (DLCO) > 30% predicted, and absence of O2 requirements. For children that are not able to cooperate with pulmonary function tests (PFTs), a pulse oximetry with exercise should be attempted. If nether test can be obtained it should be clearly stated in the physician's note.
  * Liver: Transaminases < 5 x upper limit of normal and bilirubin < 3 x upper limit of normal
  * Renal: serum creatinine < 2.0 mg/dl (adults) or glomerular filtration rate (GFR) >40 mL/min/1.73m2 (peds). Patients with a creatinine > 1.2 mg/dl or a history of renal dysfunction must have glomerular filtration rate (GFR) > 40 mL/min/1.73m2.
  * Adequate performance status is defined as Karnofsky score ≥ 60% (> 16 years of age) or Lansky score ≥ 50 (pediatrics)
* If recent mold infection e.g. Aspergillus - must have minimum of 30 days of appropriate treatment before bone marrow transplant (BMT) and infection controlled and be cleared by Infectious Disease.
* Second BMT: Must be > 3 months after prior myeloablative transplant.
* Patients must be ineligible for autologous transplantation due to prior autologous transplant, an inadequate autologous stem cell harvest, inability to withstand a myeloablative preparative regimen, or clinically aggressive/high risk disease.
* Patients are eligible for transplantation if there is no evidence of progressive disease by imaging modalities or biopsy. Persistent PET activity, though possibly related to lymphoma, is not an exclusion criterion in the absence of CT changes indicating progression.
* Patients with stable disease are eligible for transplantation if the largest residual nodal mass is < 5 cm (approximately). For patients who have responded to preceding therapy, the largest residual mass must represent a 50% reduction and be < 7.5 cm (approximately).
* Voluntary written consent (adult or parental/guardian)

Exclusion Criteria:

* Available and clinically suitable 5-6/6 HLA-A, B, DRB1 matched sibling donor
* Pregnant or breastfeeding
* Evidence of HIV infection or known HIV positive serology
* Current active serious infection
* Unless in post-chemotherapy and radioimmunoconjugated antibody induced aplasia, when he/she would be eligible, patients with acute leukemia in morphologic relapse/ persistent disease defined as > 5% blasts in normocellular bone marrow OR any % blasts if blasts have unique morphologic markers (e.g. Auer rods) or associated cytogenetic markers that allows morphologic relapse to be distinguished are not eligible.
* Chronic myeloid leukemia (CML) in refractory blast crisis
* Large cell lymphoma, mantle cell lymphoma and Hodgkin disease that is progressive on salvage therapy. Stable disease is acceptable to move forward provided it is non-bulky.
* active central nervous system malignancy

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Brunstein, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Haploidentical Stem Cell Transplant: This is a treatment guideline for HLA-Haploidentical hematopoietic stem cell transplant (HSCT) using a reduced intensity conditioning (RIC) regimen. This regimen consists of fludarabine, cyclophosphamide and low dose total body irradiation (TBI).
  Fludarabine: Fludarabine 30 mg/m2 IV over 30-60 minutes on days -6 through -2 before transplant.
  Cyclophosphamide: Cyclophosphamide 14.5 mg/kg IV over 1-2 hours on days -6 and -5 before transplant and Cyclophosphamide 50 mg/kg IV on days 3 and 4 post-transplant.
  Total Body Irradiation: TBI 200cGy (centigray) on day -1 before transplant.
  Haploidentical stem cell transplant: Non-T-cell depleted bone marrow infusion
Period: Overall Study
Arm/Group | Haploidentical Stem Cell Transplant
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Haploidentical Stem Cell Transplant
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: 2 Year Survival
Description: Percentage of patients that survive 2 years post-transplant
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Haploidentical Stem Cell Transplant
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Number of Patients With Hematopoietic Engraftment
Description: Engraftment is defined as absolute neutrophil count (ANC) ≥ 5 X 10^8/L for 3 consecutive measurements.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Haploidentical Stem Cell Transplant
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Number of Patients With Chimerism
Description: Number of patients with chimerism at day 100, 6 months and 1 year
Time Frame: 100 days
Population: Chimerism at 6 months and 1 year not evaluated
Measure: Count of Participants; unit: Participants
Arm/Group | Haploidentical Stem Cell Transplant
Number analyzed (Participants) | 2
Participants
  Chimerism at day 100 | 2
  Chimerism at 6 months | NA — Data not available due to patient's death
  Chimerism at 1 year | NA — Data not available due to patient's death

4. Secondary Outcome: Number of Patients Experiencing Acute Graft-versus-host Disease by 100 Days
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Haploidentical Stem Cell Transplant
Number analyzed (Participants) | 2
Participants | 1

5. Secondary Outcome: Number of Patients Experiencing Chronic Graft-versus-host Disease by 1 Year
Time Frame: 1 year
Population: Data were not collected for this Outcome Measure as both participants died by the 6 month time point
Arm/Group | Haploidentical Stem Cell Transplant
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Patients Experiencing Transplant Related Mortality (TRM)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Haploidentical Stem Cell Transplant
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Time Frame: 2 years post-transplant
Arm/Group | Haploidentical Stem Cell Transplant
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT02145039/Prot_SAP_000.pdf